CLINICAL TRIAL: NCT02557568
Title: Evaluation of an Algorithm for Identifying Persistent Nasal Staphylococcus Aureus Carriage in a Cohort of Healthy Volunteers and Patients Regularly Monitored at the CHU of Saint-Etienne
Acronym: ScreenStaph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1108059
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Staphylococcal Infections
Keywords: nasal carriage; Staphylococcus aureus; hemodialysis patients
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemodialysis patients (HPs) (Experimental): staphylococcus aureus carriage is measured in nose
  Interventions: Other: Staphylococcus aureus carriage
- Healthcare Workers (HCWs) (Experimental): staphylococcus aureus carriage is measured in nose
  Interventions: Other: Staphylococcus aureus carriage

INTERVENTIONS:
Other: Staphylococcus aureus carriage — Staphylococcus aureus carriage is measured in the nose. Nasal samples were taken by the nursing staff of the ward using nylon flocked swab. Prior taking the sample, swabs were wetted using an additional tube containing a sponge impregnated with normal saline solution.

SUMMARY:
The nasal carriage of Staphylococcus aureus is a major risk factor of S. aureus infection, notably in hemodialysis patients (HPs). Decolonization strategies were shown able to reduce the rate of S. aureus infection in this category of patients although the risk of emergence of antimicrobial resistance persists. Approximately one quarter of the general population is colonized by S. aureus in the anterior part of the nostril (vestibulum nasi). Three main categories of nasal carriers have been historically identified: persistent carriers (20%, 12-30%]), intermittent carriers (30%, [16-70%]) and non-carriers (50% [16-69%]). By contrast to intermittent carriers and non-carriers, persistent nasal carriers have a higher risk of S. aureus infection, especially in continuous peritoneal dialysis and in orthopedic surgery.

Persistent carriers are characterized by a higher nasal bacterial load, a longer duration of carriage, a lower rate of exchange of S. aureus strains, and a particular affinity for the carried strain. However, there is no consensual definition of this persistent carriage state. In previous studies, 5 to 12 nasal sampling episodes were realized for a period ranging from 5 weeks to 8 years. The index of carriage, corresponding to the number of samples positive for S. aureus divided by the total number of samples, has been proposed to standardize the definition of the carriage state. According to standard tools, it is almost impossible to determine the nasal carriage state in routine practice.

Recently, an algorithm based on one or two quantitative cultures from nasal samples taken within 2 days that was able to distinguish accurately persistent and non-persistent nasal carriers of S. aureus has been described; only one nasal sample was needed in more than 9 cases out of 10. The aim of the present study was to assess prospectively the reliability of this algorithm in clinical practice in a cohort of healthcare workers (HCWs) and HPs and to check its ability for identifying patients with the highest risk of S. aureus infection

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers or hemodialysis patients
* carrier state of S. aureus unknown
* written consent

Exclusion Criteria:

* chronic soft skin tissue infection due to S. aureus or eczema,
* ongoing or completed antibiotic treatment for less than 15 days,
* nasal decolonization by mupirocin or skin decolonization by antiseptic bath for at least 5 consecutive days in the previous year,
* pregnancy,
* HIV infection
* hemostasis disorder.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
S. aureus nasal carriage state | 10-week period
  HPs and HCWs were sampled over a 10-week period using at least 7 and at most 12 sampling episodes. S. aureus persistent nasal carriers were defined by an index of carriage greater than or equal to 0.8 and S. aureus intermittent nasal carriers by a positive index of carriage lower than 0.8. An index of carriage is defined for each patients by the ratio : positive sample/total sample

CONTACTS AND LOCATIONS:
Overall Officials: Florence Grattard, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France